CLINICAL TRIAL: NCT02662868
Title: Metastatic Breast Cancer in Brazil: Characterization of Patients and Treatments
Status: Completed | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: LACOG 0312
Record Dates: First submitted 2016-01-15; First posted 2016-01-26 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer; Metastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to describe demographics and socioeconomics characteristics associated to the diagnosis of metastatic breast cancer in Brazil.

DETAILED DESCRIPTION:
The primary aim of this study is to characterize patients and treatments of metastatic breast cancer in Brazil. Other specific aims are:

* to describe patients demographics and socioeconomic characteristics
* to describe the BC pathological characterization
* to describe treatment (describe each treatment with dates start-end, cycles, dosing, sequence and line of treatment, reason for discontinuation)
* to analyze patients outcome (time to progression, site of metastasis, progression free survival (PFS), overall survival (OS), skeletal related events (SRE))

ELIGIBILITY:
Inclusion Criteria:

* Women > 18 years old
* Patients diagnosed with de novo or recurrent metastatic breast cancer during the period of January to December 2012
* Any invasive breast cancer histology and subtype

Exclusion Criteria:

* Male breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women >18 years old, patients diagnosed with metastatic breast cancer in the year of 2012 in Brazil
Sampling Method: Non-Probability Sample
Enrollment: 767 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Description of sociodemographic and socioeconomics characteristics associated to diagnostic and treatment of metastatic breast cancer in Brazil | 8 months

SECONDARY OUTCOMES:
Description of demographic characteristics of metastatic breast cancer patients | 8 months
The clinical and pathological characteristics of patients with metastatic breast cancer | 8 months
Prior treatment for breast cancer before metastatic disease | 8 months
The description of the clinical outcome of the patient diagnosed with metastatic breast cancer | 8 months
Type of treatment after the diagnosis of metastatic breast cancer | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Werutsky, MD, Study Director — Latin American Cooperative Oncology Group
Locations (24):
- Brazil (24):
  - Centro Regional Integrado de Oncologia (CRIO), Fortaleza, Ceará
  - Hospital Haroldo Joaçaba Instituto do Câncer do Ceará, Fortaleza, Ceará
  - Clínica AMO, Salvador, Estado de Bahia
  - Clínica CEHON, Salvador, Estado de Bahia
  - Núcleo de Oncologia da Bahia - NOB, Salvador, Estado de Bahia
  - Oncovida, Brasília, Federal District
  - Instituto Nacional do Câncer, Rio de Janeiro, Rio de Janeiro
  - Hospital Tacchini, Bento Gonçalves, Rio Grande do Sul
  - CPO - Pucrs, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas em Hematologia e Oncologia, Santo André, Rio Grande do Sul
  - Centro de Pesquisas Oncológicas - CEPON, Florianópolis, Santa Catarina
  - Centro de Novos Tratamentos de Itajaí, Itajaí, Santa Catarina
  - Hospital do Câncer de Barretos, Barretos, São Paulo
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - InORP, Ribeirão Preto, São Paulo
  - Centro de Oncologia e Hematologia de Rio Claro, Rio Claro, São Paulo
  - IEP São Lucas, Santo André, São Paulo
  - Hospital AC Camargo, São Paulo, São Paulo
  - Hospital São José, São Paulo, São Paulo
  - ICESP, São Paulo, São Paulo
  - Instituto Brasileiro de Controle do Câncer - IBCC, São Paulo, São Paulo

REFERENCES:
- [Background] Edwards BK, Noone AM, Mariotto AB, Simard EP, Boscoe FP, Henley SJ, Jemal A, Cho H, Anderson RN, Kohler BA, Eheman CR, Ward EM. Annual Report to the Nation on the status of cancer, 1975-2010, featuring prevalence of comorbidity and impact on survival among persons with lung, colorectal, breast, or prostate cancer. Cancer. 2014 May 1;120(9):1290-314. doi: 10.1002/cncr.28509. Epub 2013 Dec 16. PMID 24343171
- [Background] Autier P, Boniol M, La Vecchia C, Vatten L, Gavin A, Hery C, Heanue M. Disparities in breast cancer mortality trends between 30 European countries: retrospective trend analysis of WHO mortality database. BMJ. 2010 Aug 11;341:c3620. doi: 10.1136/bmj.c3620. PMID 20702548
- [Background] Malvezzi M, Bertuccio P, Levi F, La Vecchia C, Negri E. European cancer mortality predictions for the year 2014. Ann Oncol. 2014 Aug;25(8):1650-6. doi: 10.1093/annonc/mdu138. Epub 2014 Apr 23. PMID 24759568
- [Background] Lee BL, Liedke PE, Barrios CH, Simon SD, Finkelstein DM, Goss PE. Breast cancer in Brazil: present status and future goals. Lancet Oncol. 2012 Mar;13(3):e95-e102. doi: 10.1016/S1470-2045(11)70323-0. PMID 22381937
- [Background] Liedke PE, Finkelstein DM, Szymonifka J, Barrios CH, Chavarri-Guerra Y, Bines J, Vasconcelos C, Simon SD, Goss PE. Outcomes of breast cancer in Brazil related to health care coverage: a retrospective cohort study. Cancer Epidemiol Biomarkers Prev. 2014 Jan;23(1):126-33. doi: 10.1158/1055-9965.EPI-13-0693. Epub 2013 Oct 28. PMID 24165578
- [Background] Regierer AC, Wolters R, Ufen MP, Weigel A, Novopashenny I, Kohne CH, Samonigg H, Eucker J, Possinger K, Wischnewsky MB. An internally and externally validated prognostic score for metastatic breast cancer: analysis of 2269 patients. Ann Oncol. 2014 Mar;25(3):633-638. doi: 10.1093/annonc/mdt539. Epub 2013 Dec 23. PMID 24368402
- [Background] Andre F, Neven P, Marinsek N, Zhang J, Baladi JF, Degun R, Benelli G, Saletan S, Jerusalem G. Disease management patterns for postmenopausal women in Europe with hormone-receptor-positive, human epidermal growth factor receptor-2 negative advanced breast cancer. Curr Med Res Opin. 2014 Jun;30(6):1007-16. doi: 10.1185/03007995.2014.887002. Epub 2014 Feb 3. PMID 24490834
- [Background] Baselga J, Campone M, Piccart M, Burris HA 3rd, Rugo HS, Sahmoud T, Noguchi S, Gnant M, Pritchard KI, Lebrun F, Beck JT, Ito Y, Yardley D, Deleu I, Perez A, Bachelot T, Vittori L, Xu Z, Mukhopadhyay P, Lebwohl D, Hortobagyi GN. Everolimus in postmenopausal hormone-receptor-positive advanced breast cancer. N Engl J Med. 2012 Feb 9;366(6):520-9. doi: 10.1056/NEJMoa1109653. Epub 2011 Dec 7. PMID 22149876
- [Background] Yardley DA, Noguchi S, Pritchard KI, Burris HA 3rd, Baselga J, Gnant M, Hortobagyi GN, Campone M, Pistilli B, Piccart M, Melichar B, Petrakova K, Arena FP, Erdkamp F, Harb WA, Feng W, Cahana A, Taran T, Lebwohl D, Rugo HS. Everolimus plus exemestane in postmenopausal patients with HR(+) breast cancer: BOLERO-2 final progression-free survival analysis. Adv Ther. 2013 Oct;30(10):870-84. doi: 10.1007/s12325-013-0060-1. Epub 2013 Oct 25. PMID 24158787
- [Background] Campone M, Bachelot T, Gnant M, Deleu I, Rugo HS, Pistilli B, Noguchi S, Shtivelband M, Pritchard KI, Provencher L, Burris HA 3rd, Hart L, Melichar B, Hortobagyi GN, Arena F, Baselga J, Panneerselvam A, Heniquez A, El-Hashimyt M, Taran T, Sahmoud T, Piccart M. Effect of visceral metastases on the efficacy and safety of everolimus in postmenopausal women with advanced breast cancer: subgroup analysis from the BOLERO-2 study. Eur J Cancer. 2013 Aug;49(12):2621-32. doi: 10.1016/j.ejca.2013.04.011. Epub 2013 Jun 1. PMID 23735704
- [Background] Verma S, Miles D, Gianni L, Krop IE, Welslau M, Baselga J, Pegram M, Oh DY, Dieras V, Guardino E, Fang L, Lu MW, Olsen S, Blackwell K; EMILIA Study Group. Trastuzumab emtansine for HER2-positive advanced breast cancer. N Engl J Med. 2012 Nov 8;367(19):1783-91. doi: 10.1056/NEJMoa1209124. Epub 2012 Oct 1. PMID 23020162
- [Background] Baselga J, Cortes J, Kim SB, Im SA, Hegg R, Im YH, Roman L, Pedrini JL, Pienkowski T, Knott A, Clark E, Benyunes MC, Ross G, Swain SM; CLEOPATRA Study Group. Pertuzumab plus trastuzumab plus docetaxel for metastatic breast cancer. N Engl J Med. 2012 Jan 12;366(2):109-19. doi: 10.1056/NEJMoa1113216. Epub 2011 Dec 7. PMID 22149875